CLINICAL TRIAL: NCT02490774
Title: Multi-center, Randomized, Comparator-controlled, Single-blind, Parallel-group Study to Investigate the Pharmacodynamics, Pharmacokinetics and Safety of an Intrauterine System Releasing BAY 1007626, as Compared With Mirena and Jaydess, in a Combined Proof-of-concept and Dose-finding Study in Healthy Pre Menopausal Women Treated for 90 Days
Brief Title: To Investigate the Pharmacological Effects, Drug Blood Levels and Safety of an Intrauterine System Releasing the Study Drug BAY1007626 in Comparison to Mirena and Jaydess in Healthy Young Women Treated for 90 Days to Determine the Drug Dose for Further Development
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15731; 2013-003980-74 (EudraCT Number)
Record Dates: First submitted 2015-06-02; First posted 2015-07-07 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Contraception
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm 1: BAY1007626, low relase (Experimental): Intrauterine device with a low in vitro release rate
  Interventions: Drug: BAY1007626
- Arm 2: BAY1007626, low to medium release (Experimental): Intrauterine device with a low to medium in vitro release rate
  Interventions: Drug: BAY1007626
- Arm 3: BAY1007626, medium release (Experimental): Intrauterine device with a medium in vitro release rate
  Interventions: Drug: BAY1007626
- Arm 4: BAY 1007626, high release (Experimental): Intrauterine device with a high in vitro release rate
  Interventions: Drug: BAY1007626
- Arm 5: Levonorgestrel, Jaydess (Active Comparator): Intrauterine device releasing levonorgestrel (Jaydess)
  Interventions: Drug: Jaydess
- Arm 6: Levonorgestrel, Mirena (Active Comparator): Intrauterine device releasing levonorgestrel (Mirena)
  Interventions: Drug: Mirena

INTERVENTIONS:
Drug: BAY1007626 — Intrauterine device with 4 different in vitro release rates (low, low to medium, medium, high)
  Arms: Arm 1: BAY1007626, low relase; Arm 2: BAY1007626, low to medium release; Arm 3: BAY1007626, medium release; Arm 4: BAY 1007626, high release
Drug: Jaydess — Jaydess: Intrauterine device with a nominal in vitro release of 12 µg levonorgestrel/day
  Arms: Arm 5: Levonorgestrel, Jaydess
Drug: Mirena — Mirena: Intrauterine device with a nominal in vitro release of 20 µg levonorgestrel/day
  Arms: Arm 6: Levonorgestrel, Mirena

SUMMARY:
Investigation of pharmacological effects, drug blood levels and safety of an intrauterine system releasing the study drug BAY1007626 in comparison to Mirena and Jaydess in healthy young women treated for 90 days to determine the drug dose for further development

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subject.
* Willingness to use non-hormonal methods of contraception during the study.
* This applies during the cycle preceding the pre-treatment cycle until the end of follow-up.
* Age at screening: 18-40 years inclusive.
* Body mass index (BMI) at screening: ≥ 18 and ≤ 32 kg/m².
* History of regular cyclic menstrual periods.
* No clinically relevant abnormal findings in the pre-treatment endometrial biopsy.

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal.
* Any presence or history of known or suspected malignant tumors, especially any known or suspected breast cancer or other progestin-sensitive cancer.
* Any presence or history of known or suspected benign tumors of the liver or of the pituitary or adrenal gland.
* Amenorrhea (with unknown reason, not amenorrhea due to hormonal treatment) for more than 3 months within the 6 months before the first screening examination.
* Use of short-acting preparations containing sex hormones during the cycle preceding the pre-treatment cycle (oral, transdermal, intravaginal, IUS).
* Use of long-acting preparations containing sex hormones within the 40 weeks before the first screening examination (any long-acting injectable or implant).

Clinically relevant findings in the physical examination (e.g. pronounced varicosis, thrombophlebitis, and evidence of peripheral circulatory disturbances).

Menstrual disorders with suspicion of ovarian failure (e.g., oligomenorrhea, amenorrhea, hypomenorrhea).

* Known bleeding irregularities
* Current or recurrent pelvic inflammatory disease, including pelvic inflammatory disease within 6 month prior to the insertion of the IUS and any active sexually transmitted disease.
* Anovulatory pre-treatment cycle (ovulation has to be observed by day 27 at the latest).
* Positive result of urine pregnancy test.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-07-22 (Actual)

PRIMARY OUTCOMES:
Number of bleeding and spotting days | Daily recorded during 90 days treatment period
Progestin effects on endometrial histology | Data derived from biopsies taken in the pre-treatment cycle, under treatment (between day 42 and day 90 of treatment) and during follow-up (within max. 40 days after IUS removal).
  Endometrail histology will be evaluated according to standardized criteria, derived from Blaustein's standard pathology textbook and criteria for secretory-type effects caused by exogenous progestins after intrauterine application.
Ovulation(Yes/no) | Treatment period 90 days

SECONDARY OUTCOMES:
Endometrial thickness | pre-treatment cycle days 6, 9, 12, 15, 18, 21, 24, 27, 30, treatment period days 1, 13, 27, 41, 44, 48, 51, 55, 58, 62, 65, 69, 72, 76, 79, 83, 86, 90
Bleeding characterization (Intensity, pattern) | For 90 day treatment period
  Classified using a 5-step scale from "none" to "heavy"
Serum levels of estradiol | Repeatedly under 90 day treatment
Serum levels of progesterone | Repeatedly under 90 day treatment
Serum levels of luteinizing hormone | Repeatedly under 90 day treatment
Serum levels of follicle-stimulating hormone | Repeatedly under 90 day treatment
Cervix function (Insler score) | cycle day 6,9,12,15,18,23,24,27,40, treatment period days 41,44,48,51,55,58,62,65,69,76,79,80,83,90
  The cervix function is classified using the 4-step Insler Score
Number of participants with adverse events as a measure of safety and tolerability. | up to 5 months
Cmax of BAY1007626 | treatment period days 13,20,30,41,55,62,72, 90, 91, 92,93,
AUC of BAY1007626 | treatment period days 13,20,30,41,55,62,72, 90, 91, 92,93,95
T1/2 of BAY1007626 | treatment period days 13,20,30,41,55,62,72, 90, 91, 92,93,95

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- Germany (3):
  - Hanover, Lower Saxony
  - Berlin
  - Hamburg
- Groningen, Netherlands
- Belfast, United Kingdom